CLINICAL TRIAL: NCT03555318
Title: Randomized Clinical Trial: Assessment of a Multidisciplinary Intervention by a Cardiologist and Geriatrician After Hospital Admission Due to Heart Failure in Elderly Patients.
Brief Title: Intervention by a Cardiologist and Geriatrician in Elderly Patients After Admission Due to Heart Failure.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Fundacion MAPFRE (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/7653/I
Record Dates: First submitted 2018-05-07; First posted 2018-06-13 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2019-11

CONDITIONS: Heart Failure
Keywords: Heart failure; Frailty; Outcome; Hospitalization; Mortality
MeSH Terms: conditions — Heart Failure; Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Geriatrician + Cardiologist (Experimental): Patients randomized to a combined ambulatory follow up with a cardiologist and a geriatrician.
  Interventions: Other: Combined ambulatory visit; Other: Geriatric intervention
- Cardiologist (Active Comparator): Patients randomized to usual care (ambulatory follow up with a cardiologist).
  Interventions: Other: Ambulatory visit

INTERVENTIONS:
Other: Ambulatory visit — All patients will have an ambulatory visit with the cardiologist.
  Arms: Cardiologist
Other: Combined ambulatory visit — Both the geriatrician and cardiologist will evaluate the patient and cardiac treatment will be agreed on between both specialists.
  Arms: Geriatrician + Cardiologist
Other: Geriatric intervention — After the geriatric assessment, measures to improve frailty will be started.
  Arms: Geriatrician + Cardiologist

SUMMARY:
Randomized clinical trial in which patients with a recent admission for heart failure in the cardiology department of the Hospital de Mar will be randomized to usual follow-up (cardiologist of the Heart Failure Unit) or follow-up by cardiologist and intervention by the geriatrician. This visit will be done at the same time. The main gial of this study is to evaluate whether the combined intervention of a cardiologist and a geriatrician reduces hospital all-cause rehospitalizations at 1 year.

DETAILED DESCRIPTION:
Patients will be invited to participate on the day of hospital discharge. Once the informed consent has been signed, patients will be randomized with a 1: 1 ratio to conventional follow-up (cardiologist) or combined follow-up (ambulatory visit with cardiologist and geriatrics on the same day). Randomization will be stratified according to the presence or absence of criteria of frailty and ventricular function (cut-off 50%) to ensure that both groups are balanced. This stratification will be achieved by generating 4 different randomization lists. Frailty will be assessed using the Canadian Study of Health and Aging (CSHA) Clinical Frailty Scale. Randomization will be carried out by administrative staff independent of the study following a computer generated randomization scheme.The first visit will be made in less than 10 days after discharge from the hospital. Lawton and Barthel index and Pfeiffer test and quality of life test will be done in both groups.

The cost associated with care in the hospital is collected in each patient and therefore the total cost of the admissions, ambulatory visits and emergencies of each patient will be retrospectively evaluated.

In patients in the intervention arm the following areas will be evaluated: social sphere (Social and family evaluation scale of Gijón (abbreviated and modified) (Barcelona version), functional capacity (Barthel index and Lawton index), cognitive sphere (Pfeiffer test), emotional sphere (Geriatric Depression Scale Yesavage), nutritional status (Mini-Nutritional Assessment Short Form, plasma albumin), comorbidity (Charlson index) and the presence of geriatric syndromes (falls, polypharmacy, ulcers pressure, constipation, incontinence, insomnia.) Interdisciplinary interventions will be carried out in each of the areas evaluated.

Follow-up will be carried out at the heart failure clinic of the Cardiology Department at 3, 6 and 12 months. A clinical event evaluation committee will be appointed, consisting of 2 independent cardiologists, who will blindly adjudicate the events that occurred during the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 75 years with a recent admission for heart failure (within the previous 10 days).

Exclusion Criteria:

* Patients in palliative care.
* Patients with chronic pathologies with expected life expectancy <1 year.
* Patients discharged to a skilled nursing facility
* Patients with heart valve replacement during index admission

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with all-cause hospitalization within the defined time points | 1 year
  Number of participants with an all-cause hospitalization at 1 year follow-up

SECONDARY OUTCOMES:
Number of participants with heart failure hospitalization within the defined time points | 1 year
  Number of participants with heart failure hospitalization at 1 year follow-up
Number of participants dead within the defined time points | 1 year
  Number of participants dead at 1 year follow-up
Change in quality of life measured with the Kansas City Cardiomyopathy Questionnaire (KCCQ) within the defined time points | 1 year
  Change in quality of life measured with the Kansas City Cardiomyopathy Questionnaire (KCCQ), a self-applicable health related quality of life instrument specific to heart failure, within the defined time points. The KCCQ ranges from 0 to 100, with 100 being the best state. A change in 5 points at 1 year follow-up will be considered clinically relevant.
Change in functional capacity measured with the Barthel index within the defined time points | 1 year
  Change in functional capacity measured with the Barthel index at 1 year follow-up
Change in the number of participants with more than 5 medications (polypharmacy) within the defined time points | 1 year
  Change in the number of participants with more than 5 medications (polypharmacy) at 1 year follow-up
Differences in total number of outpatient visits, emergency room visits and hospitalizations (resource use) within the defined time points | 1 year
  Differences in total number of outpatient visits, emergency room visits and hospitalizations (resource use) at 1 year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nuria Farre, MD, Principal Investigator — Institut Hospital del Mar d'Investigacions Mèdiques
Locations (1):
- Hospital del Mar, Parc de Salut Mar, Barcelona, Non-USA, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luiso D, Herrero-Torrus M, Badosa N, Roqueta C, Ruiz-Bustillo S, Belarte-Tornero LC, Valdivielso-More S, Morales RO, Vazquez O, Farre N. Quality of Life in Older Patients after a Heart Failure Hospitalization: Results from the SENECOR Study. J Clin Med. 2022 May 27;11(11):3035. doi: 10.3390/jcm11113035. PMID 35683423
- [Derived] Herrero-Torrus M, Badosa N, Roqueta C, Ruiz-Bustillo S, Sole-Gonzalez E, Belarte-Tornero LC, Valdivielso-More S, Vazquez O, Farre N. Randomized Controlled Trial Comparing a Multidisciplinary Intervention by a Geriatrician and a Cardiologist to Usual Care after a Heart Failure Hospitalization in Older Patients: The SENECOR Study. J Clin Med. 2022 Mar 30;11(7):1932. doi: 10.3390/jcm11071932. PMID 35407540